CLINICAL TRIAL: NCT06543134
Title: Evaluation of The Relationship Between Perioperative Hypothermia and Emergence Agitation
Status: Recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Aleyna Cicek, Anesthesiologist, Kocaeli City Hospital
Other Study IDs: ACicek
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Hypothermia; Anesthesia; Agitation, Emergence; Postoperative Complications; Hypothermia Following Anesthesia
Keywords: Hypothermia; Agitation; Emergence; Recovery from anesthesia; Postoperative Complications
MeSH Terms: conditions — Hypothermia; Emergence Delirium; Postoperative Complications; Psychomotor Agitation | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients who developed postoperative hypothermia were included in this group.
  Interventions: Procedure: surgery; Procedure: sedation scale
- Group B: Patients who did not develop postoperative hypothermia were included in this group.
  Interventions: Procedure: surgery; Procedure: sedation scale

INTERVENTIONS:
Procedure: surgery — ENT surgery lasting more than half an hour
Procedure: sedation scale — Measurement of postoperative recovery with the Richmond agitation scale and the Riker sedation scale

SUMMARY:
The main aim of our study was to investigate the relationship between perioperative hypothermia and postoperative emergence agitation.

DETAILED DESCRIPTION:
Unintentional hypothermia during surgery is defined as a decrease in body temperature below 36.0 C in the preoperative period, 1 hour before anesthesia and within the first 24 hours after surgery (1).

Unintentional hypothermia during surgery is seen in most patients undergoing surgery. The incidence of perioperative hypothermia is expressed with different values in different studies, but it varies between 30% and 90% (2,3). Hypothermia has many negative effects on mortality and morbidity, such as increased hospital stay, increased perioperative bleeding, increased cardiac complications, delayed wound healing, and delayed recovery from anesthesia (4). It has been observed that these negative effects are seen even in mild hypothermia and that patients should take a more active role in preventing perioperative hypothermia (5). Risk factors for perioperative hypothermia include many factors such as prolonged surgery, advanced age, ASA score, gender, and intravenous fluid administration.

The mentioned negative situation is a negative situation. Recovery agitation was first described in the 1960s and is characterized by restlessness, crying, and poor cooperation (6). Recovery agitation may be severe in the first 30 minutes and then subside. During this time, it may lead to self-harm, disruption of surgical drains or dressings, increased bleeding and surgical complications, unintended early extubations, and an increase in falls and other similar complications in patients (7). Recovery agitation in pediatric patients is measured by the Pediatric Anesthesia Early Delirium Scale and in adult patients, usually by the Richmond Agitation Sedation Scale (8). The incidence of recovery agitation is approximately 20%, and its pathophysiology is not yet fully understood. Risk factors include age, gender, ASA physical status, type of surgery, anesthetic technique (inhalation or total intravenous), administration of neostigmine or doxapram, inadequate postoperative analgesia, pain, presence of a tracheal tube, and presence of a urinary catheter (9). In our literature review, we observed that the effects of perioperative hypothermia and core temperature changes on recovery agitation have not been sufficiently investigated. In this study, we aimed to investigate the relationship between perioperative hypothermia and recovery agitation in patients undergoing septoplasty/rhinoplasty, functional endoscopic sinus surgery (FESS), tympanoplasty, and mastoidectomy in otolaryngology operating rooms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with informed consent Elective planned cases
* Patients between the ages of 18-65
* American Society of Anesthesiologists ASA classification ASA 1-2 patients
* Surgeries planned to last at least 30 minutes.

Exclusion Criteria:

* Patients who refuse to participate in the study,
* patients who are considered for emergency surgery,
* pediatric patients,
* patients with peripheral vascular diseases or carotid stenosis,
* patients using antidepressants or antipsychotic drugs
* those with neurological diseases will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will be operated in ENT operating rooms in a tertiary education and research hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Relationship between hypothermia and emergence agitation | first postoperative hour
  Comparison of recovery agitation rates in postoperative hypothermic and non-hypothermic patients

SECONDARY OUTCOMES:
Incidence of perioperative hypothermia | Between the first 1 hour preoperatively and the first 1 hour postoperatively
  Incidence of hypothermia observed in the operating room and recovery room

OTHER OUTCOMES:
Comparison of agitation/sedation rates in hypothermic patients | Between the first 1 hour preoperatively and the first 1 hour postoperatively
  Comparison of agitation/sedation rates in hypothermic patients will be compared by measuring percentages

CONTACTS AND LOCATIONS:
Overall Officials: Aleyna Çiçek, md, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient data can be obtained from the health directorate with appropriate permission and request. Data collected for research will not be shared.

REFERENCES:
- [Background] Yu D, Chai W, Sun X, Yao L. Emergence agitation in adults: risk factors in 2,000 patients. Can J Anaesth. 2010 Sep;57(9):843-8. doi: 10.1007/s12630-010-9338-9. Epub 2010 Jun 5. PMID 20526708
- [Background] Demir CY, Yuzkat N. Prevention of Emergence Agitation with Ketamine in Rhinoplasty. Aesthetic Plast Surg. 2018 Jun;42(3):847-853. doi: 10.1007/s00266-018-1103-4. Epub 2018 Feb 20. PMID 29464385
- [Background] Chen L, Xu M, Li GY, Cai WX, Zhou JX. Incidence, Risk Factors and Consequences of Emergence Agitation in Adult Patients after Elective Craniotomy for Brain Tumor: A Prospective Cohort Study. PLoS One. 2014 Dec 10;9(12):e114239. doi: 10.1371/journal.pone.0114239. eCollection 2014. PMID 25493435
- [Background] Lee SJ, Sung TY. Emergence agitation: current knowledge and unresolved questions. Korean J Anesthesiol. 2020 Dec;73(6):471-485. doi: 10.4097/kja.20097. Epub 2020 Mar 25. PMID 32209961